CLINICAL TRIAL: NCT02444572
Title: Comparison of Thromboembolic Events in Patients Undergoing Gastrointestinal Cancer Surgery and Thromboprophylactic Treatment With Two Enoxaparin Formulations (ENOXA® vs Lovenox®)
Brief Title: Comparison of Thromboembolic Events in Patients Undergoing Thromboprophylactic Treatment With ENOXA® vs Lovenox®
Acronym: ENOXACARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ENOXACARE_med14
Record Dates: First submitted 2015-05-07; First posted 2015-05-14 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Gastrointestinal Neoplasms; Thromboembolic Event
Keywords: Enoxaparin; Immunogenicity
MeSH Terms: conditions — Gastrointestinal Neoplasms; Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ENOXA® group (Experimental): Patients under ENOXA® 4000 IU according to randomization:
  * Administer ENOXA® 4000 IU (Enoxaparin 4000 IU) per day, regardless of the patient's weight at inclusion
  * Start injections 12 hours after the surgical procedure
  * Administer ENOXA® subcutaneously
  * The administration of ENOXA® should be at the same time on a daily basis for 30 successive days as per the american and french clinical guidelines
  Interventions: Drug: Enoxaparin 4000 IU
- LOVENOX® group (Active Comparator): Patients under LOVENOX® 4000 IU according to randomization:
  * Administer LOVENOX® 4000 IU (Enoxaparin 4000 IU) per day, regardless of the patient's weight at inclusion
  * Start injections 12 hours after the surgical procedure
  * Administer LOVENOX® subcutaneously
  * The administration of LOVENOX® should be at the same time on a daily basis for 30 successive days as per the american and french clinical guidelines
  Interventions: Drug: Enoxaparin 4000 IU

INTERVENTIONS:
Drug: Enoxaparin 4000 IU
  Other Names: ENOXA®; LOVENOX®

SUMMARY:
Prospective, monocentric, randomized, parallel group, rater-blinded study using two formulations of Enoxaparin sodium (ENOXA® vs LOVENOX®) to compare the thromboembolic events (symptomatic and asymptomatic) in patients undergoing gastrointestinal cancer surgery and thromboprophylactic treatment with either Enoxaparin formulations.

The study has a secondary focus as to evaluate the immunogenicity of the two formulations of Enoxaparin through a subgroup analysis.

Study followup duration is up to 30 days post surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years
* Gastrointestinal (GI) Cancer
* Elective or emergency surgery
* Preventive administration of enoxaparin sodium

Exclusion Criteria:

* Patients participating in another study
* Unfractionated heparin (UFH) use up to 30 days prior to surgical procedure
* Renal failure with creatinine clearance <30 ml / min
* Known history of peripheral venous thrombosis and/or deep venous thrombosis in the 3 months prior to inclusion
* Pregnant or breastfeeding women or women of childbearing age not using medically accepted contraceptive method
* Anticoagulant use in the 3 months prior to inclusion
* Patients with known haemostatic disorder
* Patients not consenting to participate in the study, or not capable of understanding its objectives

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Incidence of asymptomatic Deep Venous Thrombosis (DVT) | 7 - 10 days postoperative
  To compare the incidence of asymptomatic DVT, assessed by Echo Doppler of the lower limbs, between the two study treatment arms

SECONDARY OUTCOMES:
Incidence of symptomatic thromboembolic events | 30 days postoperative
  Compare the incidence of symptomatic DVT and pulmonary embolism (PE) between the two study treatment arms
Number of adverse events | 30 days postoperative
  To compare the safety of both the study of products
Incidence of both Enoxaparin formulations immunogenicity | 0 -10 days postoperative
  To compare the levels of platelet factor 4 (PF4)-Heparin complex antibodies an platelet count between the two study treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Chadli DZIRI, MD, Principal Investigator — Charles Nicolle Hospital
Locations (1):
- Charles Nicolle Hospital, Tunis, Tunis BAB Souika, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dziri C, Ben Hmida W, Dougaz W, Khalfallah M, Samaali I, Jerraya H, Bouasker I, Nouira R. Biosimilar versus branded enoxaparin to prevent postoperative venous thromboembolism after surgery for digestive tract cancer: Randomized trial. PLoS One. 2023 Nov 1;18(11):e0293269. doi: 10.1371/journal.pone.0293269. eCollection 2023. PMID 37910523